CLINICAL TRIAL: NCT06748911
Title: Use of a Detachable String Capsule for Evaluation of Barrett's Esophagus
Brief Title: Navicam for Detection of Barrett's Esophagus
Acronym: DS-MCE-BE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Swathi Eluri, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 24-000150
Record Dates: First submitted 2024-12-10; First posted 2024-12-27 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Long Segment Barrett's Esophagus (LSBE) (Experimental): Subjects diagnosed with Long Segment Barrett's Esophagus (LSBE)
  Interventions: Device: NaviCam Detachable String Capsule
- Short Segment Barrett's Esophagus (SSBE) (Experimental): Subjects diagnosed with Short Segment Barrett's Esophagus (SSBE)
  Interventions: Device: NaviCam Detachable String Capsule
- Gastro Esophageal Reflux Disease (Experimental): Subjects with Gastro Esophageal Reflux Disease (GERD) who are eligible for Barrett's Esophagus screening
  Interventions: Device: NaviCam Detachable String Capsule

INTERVENTIONS:
Device: NaviCam Detachable String Capsule — Subjects will swallow the NaviCam capsule with 20 ml water while positioned in the upright position. Once the capsule reaches the gastric cardia, the string will slowly be pulled up to systematically inspect the Z-line and upper, middle, and lower thirds of the esophagus guided by real-time viewing and by moving the capsule solely with the tether. Images will be captured at a rate of 2 frames per second.

SUMMARY:
Using a non-invasive capsule system to achieve optimal viewing angles of the esophagus for detection of Barrett's esophagus

ELIGIBILITY:
Inclusion Criteria

* Adults greater than or equal to 22 years of age with or without Barrett's Esophagus
* All Patients:

  o Have had an endoscopy within 1 year of baseline enrollment
* Patients with Barrett's Esophagus:

  * Presence of at least 1cm of salmon colored mucosa with corresponding biopsies showing intestinal metaplasia who are treatment naïve and undergoing surveillance Or
  * Chronic Gastro Esophageal Reflux Disease (GERD) patients with at least 3 additional risk factors that meet Barrett's Esophagus screening criteria per latest clinical guidelines

Exclusion Criteria

* Inability to comprehend or read the consent form
* Have an oropharynx, esophageal, or gastro-esophageal tumor
* Ongoing symptoms of dysphagia
* Presence of active clinically significant stricture
* History of stricture requiring dilation
* Presence of pacemaker or implanted cardiac defibrillator
* History of esophageal surgery with the exception of fundoplication
* Pregnancy
* History of surgery or obstructive process of the small bowel
* BMI > 38

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Detection of Columnar lined epithelium in the esophagus | From start of procedure to removal of capsule, assessed up to 30 minutes timeframe from start to end of procedure..
  Detection of Columnar lined epithelium in the esophagus

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | 30 minutes post-procedure
  Visual Analogue Scale (VAS) is an 11-tem questionnaire assessing pain, where 0 represents the "worst experience" and 10 the "best experience". Total scores range from 0 - 110, lower scores indicating lower pain and higher scores indicating greater pain.
Spielberger State-Trait Anxiety Inventory (STAI-6) | Baseline, 30 minutes post-procedure
  Patient anxiety will be measured using the shorter 6 item form of the Spielberger State-Trait Anxiety Inventory (STAI-6), with a score over 40 as a threshold for clinically significant anxiety
Impact of Events Scale (IES) | Baseline, 7 days post-procedure
  The Impact of Events Scale (IES) will be used to assess distress associated with the procedure and procedure acceptability. The IES is rated on a scale of 0 (not at all) to 4 (extremely), with higher scores indicating a greater level of distress.

CONTACTS AND LOCATIONS:
Overall Officials: Swathi Eluri, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No